CLINICAL TRIAL: NCT03382808
Title: Emotion Recognition Training in Antisocial Violent Offenders With Psychopathic Traits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCHO 1448/3-1
Record Dates: First submitted 2017-12-12; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Psychopathy; Violent Aggressive Behavior; Emotional Problem
MeSH Terms: conditions — Antisocial Personality Disorder; Aggression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEE Training (Experimental): The training sequence comprises four weekly sessions using a modified dote-probe paradigm (fearful vs. neutral expression).
  Interventions: Behavioral: SEE Training
- GAZE Training (Active Comparator): The GAZE training sequence comprises four weekly sessions using a modified dote-probe paradigm (averted vs. directed gaze).
  Interventions: Behavioral: GAZE Training

INTERVENTIONS:
Behavioral: SEE Training — Participants are first presented with a fixation cross which indicates the beginning of a trial and is immediately followed by a bilateral presentation of a neutral and a fearful image (face) of the same model identity. The fearful expression is always replaced by an arrow pointing to the left or the right which remaines active until the participant indicates via button-press which direction the arrow is pointing to. The model identity, the position of the fearful cue and the arrow probe direction are pseudo-randomized across trials with no more than three identical sequential occurrences on each parameter. Each session consists of 360 trials in total, with 120 distinct trial types and three repetitions. Participants are trained with neutral and 75% fearful expressions only in the first session; the intensity of the fearful cue is successively decreased by 15% at every subsequent session.
  Arms: SEE Training
Behavioral: GAZE Training — Participants are first presented with a fixation cross, which indicates the beginning of a trial and is immediately followed by a bilateral presentation of a direct gaze-image (neutral face) and an image of a neutral face (same model identity) displaying deviated gaze. The averted gaze-face is always replaced by an arrow pointing to the left or the right which remaines active until the participant indicates via button-press which direction the arrow is pointing to. The model identity, the position of the fearful cue and the arrow probe direction are pseudo-randomized across trials with no more than three identical sequential occurrences on each parameter. Each session consists of 360 trials in total, with 120 distinct trial types and three repetitions. Participants are trained with direct and 100% averted gaze images only in the first session; the intensity of the deviated gaze cue is successively decreased by 20% at every subsequent session.
  Arms: GAZE Training

SUMMARY:
Impaired recognition of affective facial expressions has been conclusively linked to antisocial and psychopathy. However, little is known about the modifiability of this deficit. This study aims to investigate whether and under which circumstances the proposed perceptual insensitivity can be addressed with a brief implicit training approach.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ASPD diagnosis
* PCL-Score available
* arrested for committing violent crimes

Exclusion Criteria:

* Insufficient knowledge of the German language
* Diagnosed with schizophrenia
* Substance abuse
* Neurological disease (e.g. epilepsy)
* Mental retardation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Animated morph task | change from pre-treatment to post-treatment after 8 weeks
  Morphed images are presented, beginning with the neutral face that progresses into one of the six affective expressions. This procedure creates the impression of an animated clip depicting the development of facial emotive expressions. Participants are instructed to press a button as soon as they are able to identify the emerging expression.

SECONDARY OUTCOMES:
Unconscious processing of affective facial expressions during interocular suppression in a breaking Continuous flash suppression paradigm | pre-treatment, after 8 weeks (post-treatment)
  Change in processing of unaware/unconsciously perceived emotional stimuli as assessed by number of faces correctly identified
Eye-Tracking | pre-treatment, after 8 weeks (post-treatment)
  Change in recognition and visual processing of emotional faces as indicated by raw scores and group means for dwell time, total dwell time, and time to first AOI (mouth/eye region) hit
Ambivalence Task | pre-treatment, after 8 weeks (post-treatment)
  Change in interpretation of ambiguous emotional faces as indicated by number of hostile judgments
Emotional search paradigm | pre-treatment, after 8 weeks (post-treatment)
  Assessment of implicit perceptual biases for and explicit categorization of facial expression in an emotional search paradigm (change pre- to post-intervention)
Affective prosody | pre-treatment, after 8 weeks (post-treatment)
  Change in recognition of non-verbal emotional aspects of language as assessed by number of correct classifications
Multifaceted empathy test | pre-treatment, after 8 weeks (post-treatment)
  Assessment of cognitive and emotional empathy (change pre- to post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schönenberg, PhD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tübingen, Tübingen, Baden Würrtemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schonenberg M, Christian S, Gausser AK, Mayer SV, Hautzinger M, Jusyte A. Addressing perceptual insensitivity to facial affect in violent offenders: first evidence for the efficacy of a novel implicit training approach. Psychol Med. 2014 Apr;44(5):1043-52. doi: 10.1017/S0033291713001517. Epub 2013 Jul 1. PMID 23809680
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104